CLINICAL TRIAL: NCT04681690
Title: German National Registry for Nephron-Sparing Surgery
Brief Title: German National Registry for NSS
Status: Recruiting | Type: Observational
Sponsor: Association of Urologic Oncology (AUO) (Other)
Collaborators: IAG-N at German Cancer Association (Deutsche Krebsgesellschaft e. V.) (Unknown)
Responsible Party: Sponsor
Other Study IDs: G-NeSS
Record Dates: First submitted 2020-09-09; First posted 2020-12-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Kidney Neoplasm
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, observation only. — Observation only

SUMMARY:
The G-NeSS Registry prospectively collects data on clinical and outcome variables from patients undergoing partial nephrectomy for renal masses. Analyses of data aims at identifying key factors determining the quality of surgical care in this patient population.

DETAILED DESCRIPTION:
Today the majority of patients with renal tumors is diagnosed with localized disease amenable to nephron-sparing surgery (NSS). Partial nephrectomy (PN) constitutes the reference standard treatment for small renal masses according to international guidelines. Open PN ist still the predominant apporach in Germany, but the use of minimally-invasive surgery has continously increased over the last decades. Specifically, robotic surgery is on the rise and may facilitate the adoption of a minimally-invasive PN approach even in more complex renal tumours. Real world data on the outcomes of PN according to the surgical approach are limited. Data from cancer registries and health insurance databases usually lack important information an key patient und tumour characteristics, such as tumour complexity.

The G-NESS registry database aims at prospectively collecting such clinical and outcome data from patients undergoing PN. Data collection includes perioperative variables on patient characteristics, tumour location and complexity, surgical approach, intra-/postoperative complications, and kidney function. Follow-up based on questionnaires is conducted after predefined intervals (i.e. 30 days, 12 months, 24 months, and 60 months) in order to receive information on long-term kidney function, comorbidities, and survival. The information received from the database can help to better define the optimal surgical care for patients with renal masses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* Localized renal parenchymal mass amenable to nephron-sparing surgery
* Adequate imaging of the abdomen (CT or MR with contrast)

Exclusion Criteria:

* Patient with (or suspected to have) urothelial cancer of the kidney
* Prior nephron-sparing surgery on ipsilateral kidney
* metastasized renal cell carcinoma

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a renal mass eligible for partial nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Complication rate | 60 months
  Complication rate according to Clavien-Dindo in %
Postoperative glomerular inflitration rate | 60 months
  Rate in ml/min.
Survival | 60 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Nina Harke, Dr., Study Chair — MHH; Stefan Siemer, Prof. Dr., Study Chair — University Saarland; Steffen Weikert, Prof. Dr., Study Chair — Vivantes Humboldt-Klinikum
Locations (5):
- Germany (5):
  - Sana Klinikum Hof, Hof, Bavaria
  - MHH, Hanover, Lower Saxony
  - Alexianer St. Hedwig-Krankenhaus, Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - Saarland University, Homburg/Saar